CLINICAL TRIAL: NCT01542060
Title: A Clinical Experience Programme to Collect Data on the Safety and Efficacy of NovoMix® 30 in the Treatment of Patients With Type 2 Diabetes in Jordan
Brief Title: Efficacy and Safety of Biphasic Insulin Aspart 30 for the Treatment of Type 2 Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Public Access to Clinical Trials, Novo Nordisk A/S
Other Study IDs: BIASP-1892
Record Dates: First submitted 2012-02-15; First posted 2012-03-01 (Estimated); Last update posted 2012-04-12 (Estimated); Status verified 2012-04

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- BIAsp 30 users
  Interventions: Drug: biphasic insulin aspart 30

INTERVENTIONS:
Drug: biphasic insulin aspart 30 — Administered via an insulin injection device. Dosages varied according to individual patients' medical requirement as determined by their attending clinician

SUMMARY:
This study is conducted in Asia. The aim of this observational study is to collect efficacy and safety data of biphasic insulin aspart (NovoMix® 30) in type 2 diabetes under normal clinical practice conditions.

ELIGIBILITY:
Inclusion Criteria:

* Subjects from hospitals or clinics, diagnosed with type 2 diabetes mellitus

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients from hospitals or clinics diagnosed with type 2 diabetes mellitus
Sampling Method: Non-Probability Sample
Enrollment: 298 (Actual)
Dates: Start 2004-01; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
HbA1c (glycosylated haemoglobin)

SECONDARY OUTCOMES:
FBG (Fasting Blood Glucose)
Quality of life assessed through the WHO-DTSQ (World Health Organization-Diabetes Treatment Satisfaction Questionnaire)
Incidence of adverse events
Incidence of hypoglycaemic episodes

CONTACTS AND LOCATIONS:
Overall Officials: Corporate Vice President for diabetes and devices, Study Director — Novo Nordisk A/S
Locations (1):
- Amman, Jordan

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com